CLINICAL TRIAL: NCT06360146
Title: COMPARISON OF EARLY MOBILISATION EXERCISES AND TRADITIONAL PHYSIOTHERAPY FOLLOWING CARDIAC SURGERY ON OLDER PATIENTS
Brief Title: Early Mobilisation of Post Cardiac Surgery in Geriatrics.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, İSMAİL CEYLAN, Head of hand therapy clinic. PhD., Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120685123
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Disease
Keywords: early rehabilitation; geriatrics; cardiac surgery
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): The patients in early mobilization group underwent early mobilization and functional exercises program, while the patients served as the control group did not receive the therapy protocol applied in the early mobilization group
  Interventions: Other: Early mobilisation
- Group 2 (Active Comparator): The patients in early mobilization group underwent early mobilization and functional exercises program, while the patients served as the control group did not receive the therapy protocol applied in the early mobilization group
  Interventions: Other: Early mobilisation

INTERVENTIONS:
Other: Early mobilisation — Breathing exercises, inspiratory muscle strength, postural drainage, functional exercise (stand up and sitting down on the chair, walking inward, back-ward ,and sideways), weight shifts from left to right, step up inside the patch , one leg stand, squatting leaning against wall) for three times per the day and repetition fifteen times (3 times per day for 15 repetition) and supervised walking with increments of 2 minutes, as tolerated up to 6 minutes or more at the morning, afternoon, evening and at night.

SUMMARY:
Heart and blood vessel problems together referred to as cardiovascular diseases (CVD) include congenital heart disease, cerebrovascular illness, and coronary heart disease.

Following heart surgery, patients who are active in the postoperative phase stay in the hospital for shorter periods of time and experience fewer complications.

After cardiac surgery, older adults who exercise during the recovery period experience fewer difficulties and hospitalizations.

A total of 100 elderly patients-69 men and 31 women-who had undergone cardiac surgery and were up to 65 years old-voluntarily took part in the study. There were fifty patients in each of the two groups that the participants were divided into: the early mobilization group (Group A) and the control group (Group B).

Older patients undergoing cardiac surgery also experienced improved balance as a result of early mobilization and functional exercises.

DETAILED DESCRIPTION:
A total of 100 geriatric patients-69 men and 31 women-who had undergone heart surgery and were up to 65 years old-voluntarily took part in the study. There were fifty patients in each of the two groups that the participants were divided into: the early mobilization group (Group A) and the control group (Group B). The patients in early mobilization group underwent early mobilization and functional exercises program, while the patients served as the control group did not receive the therapy protocol applied in the early mobilization group

ELIGIBILITY:
Inclusion Criteria:

Individuals who had previously had valve replacement procedures or coronary artery bypass grafting (CABG) and if all of these procedures were done by sternotomy were included in the study. The study's patients were all classified as geriatric, with ages ranging from 65 to 75. There were people of both genders in the sample. Throughout their recovery, patients who were awake, conscious, and able to communicate vocally as well as those who were able to understand and complete scales and questionnaires. Patients who signed consent forms voluntarily agreed to participate, as well as those who successfully passed the two-minute walk test (2MWT), which assesses how long it takes to walk for two minutes.

Exclusion Criteria:

* Patients unable to complete the two-minute walk test (2MWT), scales, or questionnaires. Individuals who suffered from stroke, extensive bleeding, renal failure or insufficiency, atrial fibrillation, the necessity for a second operation, or a serious infection of the sternal wound following surgery. Those who struggle with vocal and auditory communication. individuals who underwent surgery and had a pacemaker inserted. those who have experienced a prior cerebrovascular accident. Those who have suffered from neurological disorders like hemiplegia after heart surgery and mental health problems like intellectual incapacity.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire | 0-7 days
  The Short Form of the International Physical Activity Questionnaire (SF-IPAQ) was used to measure physical activity (PA). Participants were asked to describe how many days they had spent performing vigorous, moderate, and walking activities over the course of the previous week, as well as the duration of those activities

SECONDARY OUTCOMES:
Two Minute Walking Test | 0-7 days
  The 2MWT was performed over a 50-ft (15.2-m) out-and-back course. Participants were instructed to walk as fast as they could until asked to stop. They were also told not to worry if they had to slow down or rest, but that if they stopped they should start walking again as soon as they felt ready to do so. When 1 minute had elapsed, they were told "You are doing well; you have 1 minute left." Participants stopped walking at 2 minutes, and the distance covered was documented

CONTACTS AND LOCATIONS:
Locations (1):
- İsmail Ceylan, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khadanga S, Savage PD, Ades PA. Resistance Training for Older Adults in Cardiac Rehabilitation. Clin Geriatr Med. 2019 Nov;35(4):459-468. doi: 10.1016/j.cger.2019.07.005. Epub 2019 Jul 3. PMID 31543178